CLINICAL TRIAL: NCT01258686
Title: A Double-blind Phase III Study With Silymarin in the Patients Infected With HCV Who Failed Conventional Antiviral Therapy
Brief Title: Clinical Study With Silymarin in the Patients With Chronic Hepatitis C Infection Who Failed Conventional Antiviral Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK SIL-C-301
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Silymarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- silymarin, treatment (Experimental)
  Interventions: Drug: Silymarin
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silymarin — 700mg thrice daily
  Arms: silymarin, treatment
Drug: Placebo — Placebo 700mg thrice daily
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of silymarin 700 mg thrice daily and assess the safety in patients with hepatitis C virus infection compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years at screening.
2. Serum HCV RNA above quantifiable level of detection after the end of previous therapy.
3. ALT > 60 IU/L (i.e., approximately 1.5 X upper limit of normal) obtained during the screening period.
4. Previous treatment with any interferon-based therapy but 1) without sustained virological response or 2) HCV RNA detected at the end of the treatment or 3) HCV RNA undetected during the treatment and detected after or 4) have partial response(HCV RNA < 2log10 but is not eradicated) or 5) have no response or 6) discontinuation due to side effect
5. Negative urine pregnancy test (for women of childbearing potential). Females of childbearing potential must be using effective contraception during the study.

Exclusion Criteria:

1. ALT ≥ 10*ULN(Upper Limit of Normal) at the screening
2. Use of silymarin or other milk thistle preparations within 30 days prior to screening.
3. Use of other antioxidants such as vitamin E, vitamin C, glutathione, alpha-tocopherol, or non-prescribed complementary alternative medications (including dietary supplements, megadose vitamins, herbal preparations, and special teas) within 30 days prior to screening. A multivitamin at standard doses will be allowed.
4. Use of silymarin or other antioxidants or non-prescribed complementary alternative medications (as above) during the screening period or patient unwilling to refrain from taking these medications through completion of the study.
5. Any antiviral therapy within 6 months prior to screening visit.
6. Known allergy/sensitivity to milk thistle or its preparations.
7. Evidence of poorly-controlled diabetes (defined as HbA1c > 8% in patients with diabetes).
8. Use of warfarin, metronidazole or acetaminophen (greater than two grams per day) within 30 days of screening.
9. Previous Radiology test(Ultrasonography, Computed tomography,Magnetic Resonance Imaging) or liver biopsy that demonstrated presence of moderate to severe steatosis or evidence of steatohepatitis.
10. Positive test for anti-HIV or HBsAg within 5 years of screening.
11. Average alcohol consumption of more than one drink or equivalent (>12 grams) per day or more than two (2) drinks on any one day over the 30 days prior to screening. Patients who met either criterion more than 30 days ago must have consumed a monthly average of 12 grams or less per day of alcohol for at least six months prior to screening.
12. History of other chronic liver disease, including metabolic diseases, documented by appropriate test(s).
13. Women with ongoing pregnancy or breast-feeding, or contemplating pregnancy.
14. Serum creatinine level 2.0 mg/dL or greater at screening or CrCl ≤ 60cc/min, or currently on dialysis. The creatinine clearance (CrCl) will be calculated according to Cockcroft-Gault.
15. Evidence of drug abuse within 6 months prior to screening or during the screening period.
16. Evidence of decompensated liver disease defined as any of the following: serum albumin <3.2 g/dl, total bilirubin > 2.0 mg/dl, or PT/INR > 1.3 times normal at screening, or history or presence of ascites or encephalopathy, or bleeding from esophageal varices.
17. History or other evidence of severe illness or any other conditions that would make the patient, in the opinion of the investigator, unsuitable for the study (such as poorly controlled psychiatric disease, coronary artery disease, or active gastrointestinal conditions that might interfere with drug absorption).
18. History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hepatitis, autoimmune hemolytic anemia, severe psoriasis, rheumatoid arthritis) that could affect inflammatory biomarkers.
19. History of solid organ or bone marrow transplantation.
20. History of thyroid disease poorly controlled on prescribed medications.
21. Use of oral steroids for more than 14 days within 30 days prior to screening.
22. Participation in a research drug trial within 6 months of enrollment.
23. Inability or unwillingness to provide informed consent or abide by the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The proportion of patient with serum ALT less than or equal to 40 IU/L or achieves at least 50% decline to less than 60 IU/L | at week 24

SECONDARY OUTCOMES:
the change from baseline in ALT and HCV RNA (log10) | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Byung Chul Yoo, MD. PhD., Principal Investigator — Samsung Medical Center
Locations (1):
- Byung Chul, Yoo, Seoul, South Korea